CLINICAL TRIAL: NCT04999748
Title: Consumer Knowledge, Attitude, and Behavior Towards Aging Skin
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: STU00215051
Record Dates: First submitted 2021-07-21; First posted 2021-08-11 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Dermatology
Keywords: Skin care, Anti-aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will conduct a cross-sectional survey from adults 18 years of age and older to examine consumer knowledge, attitudes and behavior towards aging skin.

DETAILED DESCRIPTION:
We will perform a cross-sectional survey study to understand the significance of age-related skin changes to consumers. We will recruit participants through ResearchMatch (a national free and secure online tool) and collect the following data:

Demographic information, including age, gender, race/ethnicity, geographic location, and yearly household income

* How do participants feel towards their own skin and age-related skin changes?
* Which aging-related skin changes are the most significant?
* What factors affect how participants feel towards their skin?
* What role do age-related skin changes play in other aspects of the participants' lives, such as their social and work life?
* What treatments are participants currently seeking, and what are their goals for these treatments?
* How much do they prioritize these treatments?
* What else are they hoping to do?

Using the demographic information, we will also analyze whether there are differences with:

* Age
* Gender identity
* Racial/ethnic identity
* Marital status
* Geographic location
* Yearly household income

ELIGIBILITY:
Inclusion Criteria:

* The study will include English-speaking adults (18 years or older) who voluntarily consent to participate in the survey.

Exclusion Criteria:

* Participants under the age of 18 and non-English speaking participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Open to male and female English-speaking adults(18 years or older)
Sampling Method: Non-Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency (percentage) of participants with aging-related skin concerns | 2 months
  to determine the frequency of participants who indicate having aging-related skin concerns
Frequency (percentage) of participants with social and work life impact of age-related skin changes | 2 months
  To determine the frequency of participants who indicate age-related skin changes impact their social and work life
Measure (count) the type of treatments participants are currently seeking for aging skin concerns | 2 months
  To summarize the number of participants who would prioritize certain treatments for aging skin concerns

SECONDARY OUTCOMES:
Summarize (mean/standard deviations) demographic information | 2 months
  Demographic information, including age, gender, race/ethnicity, geographic location, marital status and yearly household income will be summarize with means and standard deviations.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Fienberg School of Medicine Department of Dermatology, Chicago, Illinois, United States